CLINICAL TRIAL: NCT03252210
Title: Preoperative Stereoscopic Localization Versus Methylene Blue Localization in GGO Patients With Lung Wedge Resection:A Prospective Self-control Study.
Brief Title: Preoperative Stereoscopic Localization Versus Methylene Blue Localization in GGO Wedge Resection
Acronym: PSLVML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wen-zhao ZHONG, Deputy director of Guangdong lung cancer institute, Guangdong Provincial People's Hospital
Organization: GuangdongPPH (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PSL-1
Record Dates: First submitted 2017-08-06; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Thoracic Surgery, Video-Assisted
Keywords: Preoperative localization; Stereoscopic Localization; Wedge Resection; Ground Glass Opacity

STUDY DESIGN:
Intervention Model Description: Single group self-control study
Masking Description: Eventhough only one group of participants，different investigators perform two kinds of localization techniques.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereoscopic Versus Methylene Blue (Experimental): In the same participant,we perform both Stereoscopic and Methylene Blue localization。Then，compare the distance between the methylene blue's anchor point and the location of lesion,stereoscopic Localization's anchor point and the location of lesion,methylene blue's anchor point and stereoscopic Localization's anchor point.
  Post Hoc Multiple Comparisons
  Interventions: Procedure: Preoperative Stereoscopic Localization

INTERVENTIONS:
Procedure: Preoperative Stereoscopic Localization — 1.Confirm the nodule's location and measure the distance between the nodule and anatomic landmarks from the CT scan. 2.According to the results of the first step，confirm the needle puncture site of the chest wall. 3.After general anesthesia and Patient positioning are completed, the needle is then inserted via the needle puncture site .

SUMMARY:
This study evaluates the feasibility，accuracy and safety of Preoperative Stereoscopic Localization Versus Methylene Blue Localization in GGO Wedge Resection. In the first stage，participants will receive both Preoperative Stereoscopic Localization and Methylene Blue Localization .In the second stage,participants only receive Preoperative Stereoscopic Localization for Wedge Resection.

DETAILED DESCRIPTION:
More and more Ground Glass Opacity（GGO）are detected because of the early screening.According to Fleischner Society, for some solid GGO, surgical resection should be performed if the solid component is larger than 5mm.With the development of video-assisted thoracoscopic surgery (VATS) techniques, minimally invasive thoracic surgery has evolved considerably over the last three decades.However, localizing the small sized pulmonary nodules during VATS is challenging when there is no change in visceral pleura.

Several traditional techniques have been described to localize peripheral pulmonary nodules, including preoperative CT-guided tattooing with methylene blue, CT scan guided spiral/hook wire placement and marking with radio-opaque materials. The traditional marking method have its strong and weak points. For the strong point, It provide a credible and precise nodule location to the surgeon. For the weak points:(1)a potential risk of pneumothorax and hemothorax.(2)Methylene blue have a tendency to diffuse over a large area during surgical preparation until the nodule's location is confirmed.(3)The Preoperative localization technique would need more time for the Preoperative preparation, which would be reduce the transport's efficiency.(4)It would occupy the resource of CT's usage.(5)Some of the methods ,such as methylene blue, maybe interference with the Pathological diagnosis.(6)These methods are all invasive operation, would Cause the patients' psychological fear.

In order to avoid these weak points，the investigators use a new localization technique which has three basic steps: 1.Confirm the nodule's location in pulmonary segments. 2.Measure the distance between the nodule and anatomic landmarks on CT. 3. Estimate the changes of the distance between the nodule and anatomic landmarks after the alveolar atelectasis. The investigators have already succeed in some case.But,the further study is needed.Hence,the investigators designed a prospective study of Preoperative Stereoscopic Localization Versus Methylene Blue Localization in GGO Wedge Resection.Then,the investigators evaluate the feasibility，accuracy and safety of Preoperative Stereoscopic Localization Versus Methylene Blue Localization in GGO Wedge Resection.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative radiology revealed the solid component of GGO is larger than 5mm
2. Preoperative radiology revealed peripheral pulmonary nodule, with both size and depth less than 3 cm
3. Preoperative radiology revealed the distance from the lesion to the visceral pleura is larger than 5 mm

Exclusion Criteria:

1. Preoperative radiology revealed pneumonia or atelectasis
2. Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
3. Bleeding tendency or anticoagulant use
4. Pregnancy or breast feeding
5. Patient who can not sign permit

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-16 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
success rate of Stereoscopic Localization | 3 day
  Success localization means that the distance from lession to anchor point is less than 3.0 cm.

SECONDARY OUTCOMES:
Comparison between Stereoscopic Localization success rate and Methylene Blue Localization success rate | 3 day
  To evaluate the two kinds of Localization.Success localization means that the distance from lession to anchor point is less than 3.0 cm.
Distance from A to B | 3 day
  A:lession B：methylene blue anchor point To evaluate the accuracy of methylene blue localization.Measure the distance from lession to the methylene blue localization anchor point
Distance from A to C | 3 day
  A:lession C：Stereoscopic Localization anchor point To evaluate the accuracy of Stereoscopic Localization localization.Measure the distance from lession to the Stereoscopic Localization localization anchor point
Distance from B to C | 3 day
  B：methylene blue anchor point C：Stereoscopic Localization anchor point To evaluate the two kinds of Localization.Measure the distance from methylene blue localization anchor point to the stereoscopic localization anchor point .
The success rate of wedge resection | 3 day
  To evaluate the accuracy rate of localization
Postoperative adverse event incidence rate | 1 months
  To evaluate the incidence rate of pneumothorax or perilesional hemorrhage in participants

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Zhao Zhong, Ph.D, Principal Investigator — Guangdong Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleedehn M, Kim DH, Lee FT, Lubner MG, Robbins JB, Ziemlewicz TJ, Hinshaw JL. Preoperative Pulmonary Nodule Localization: A Comparison of Methylene Blue and Hookwire Techniques. AJR Am J Roentgenol. 2016 Dec;207(6):1334-1339. doi: 10.2214/AJR.16.16272. Epub 2016 Sep 22. PMID 27657546
- [Background] Wicky S, Mayor B, Schnyder P. Methylene blue localizations of pulmonary nodules under CT-guidance: a new procedure used before thoracoscopic resections. Int Surg. 1997 Jan-Mar;82(1):15-7. PMID 9189791
- [Background] Wicky S, Mayor B, Cuttat JF, Schnyder P. CT-guided localizations of pulmonary nodules with methylene blue injections for thoracoscopic resections. Chest. 1994 Nov;106(5):1326-8. doi: 10.1378/chest.106.5.1326. PMID 7956378